CLINICAL TRIAL: NCT03932461
Title: Vacuum Assisted Closure Versus On-demand Relaparotomy in Patients With Fecal or Diffuse Peritonitis: A Multicenter Randomized Controlled Trial
Brief Title: Vacuum Assisted Closure Versus On-demand Relaparotomy in Patients With Fecal or Diffuse Peritonitis
Acronym: VACOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Pooya Rajabaleyan, Principal investigator, Odense University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VACOR2019
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Fecal Peritonitis; Secondary Peritonitis; Diffuse; Peritonitis
MeSH Terms: conditions — Peritonitis | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Multicentre randomized non-blinded clinical trial comprising of > 4 centres. In total there will be included 320 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vacuum assisted closure (Active Comparator): The VAC® Abdominal Dressing System (KCI Vacuum Assisted Closure, San Antonio, TX, USA) will be used. Intestines, including lateral aspects, are covered by the visceral protective layer. The first layer of foam is placed in the laparostoma on the visceral protective layer and must extend below the fascia at a distance of 5 cm from the facial opening. Above this, a minimum of one piece of foam is folded and placed in the laparostoma. Finally, the laparostoma will be covered by the occlusive drape. A circular opening of approximately 5 cm in diameter will be created in the drape where the connection tubes to the vacuum pump will be placed. Simultaneously while applying the negative pressure of 125 mmHg, the wound edges are approximated manually towards the midline. Each dressing change must be performed in the operation theatre with the patient in general anesthesia and muscle relaxation.
  Interventions: Procedure: Vacuum assisted closure
- Relaparotomy "on-demand" (Active Comparator): The Isreaelsson principle includes a running suture of the fascia with a distance of 5 mm between the stitches of 5 mm and the distance to the facial edge of 5-10 mm. Monofilament PDS 2-0 or equivalent is used. The suturing is started cranially and caudally, and the sutures are tied with self-locking knots. Four times as much suture material as the length of the wound must be used. The peritoneal fluid must be cultured at closure.
  The treating surgeon decides to perform a ROD and should be guided by the patient's general condition, gastrointestinal function, renal function, and inflammatory parameters at daily rounds.
  Interventions: Procedure: Relaparotomy "on demand"

INTERVENTIONS:
Procedure: Vacuum assisted closure — The Vacuum assisted closure system consists of an abdominal dressing covering the intra abdominal viscera over the dressing there will be placed a blue sponge which will be covered by drape and connected to a vacuum pump.
  Other Names: VAC® Abdominal Dressing System, KCI, (San Antonio, TX)
  Arms: Vacuum assisted closure
Procedure: Relaparotomy "on demand" — Abdomen is closed at the index operation after source of peritonitis is treated. Every 48-hours the patients are evaluated for the need of relaparotomy based on clinical and paraclinical parameters.
  Arms: Relaparotomy "on-demand"

SUMMARY:
Multicenter randomized controlled trial including patients with fecal or diffuse peritonitis to either vacuum assisted closure or relaparotomy "on-demand".

DETAILED DESCRIPTION:
Multicenter randomized controlled trial including patients with fecal or diffuse peritonitis* to either vacuum assisted closure or relaparotomy "on-demand". The aim with our study is to compare the postoperative complications between vacuum assisted closure and relaparotomy "on-demand".

Primary endpoint is to compare peritonitis related complications and Comprehensive Complication Index (CCI) between NPWT treatment (VAC) and conventional treatment (ROD) at 30, 90 days and 1 year.

Secondary outcome parameters are: Mortality at 30, 90 days and 1 year, SOFA score and C-reactive protein measured the first seven days after index laparatomy, quality of life after 3 and 12 months (SF-36 questionnaire), ventral hernia after 3 and 12 months. (assessed by CT) and, hospital care utility within three months after index surgery. A power calculation was made which concluded that 340 patients should be included.

*Diffuse fecal peritonitis is defined as contamination of 2 out of the 4 abdominal quadrants with fecal contamination starting from the small intestine, colon or rectum.

Design

A multicenter non-blinded superiority randomized controlled trial on VAC vs. ROD. Danish, as well as other European centers, will be invited to participate

All patients over 18 with suspected diffuse peritonitis caused by perforation of the small intestine, colon or rectum with contamination in minimum 2 out of 4 abdominal quadrants, will be included.

Exclusion criteria are;

* Diffuse peritonitis originating from a different focus than the small intestine, colon or rectum
* Diffuse peritonitis originating from a perforation on the stomach, duodenum, gallbladder, appendix, necrotizing pancreatitis, salpingitis, or peritoneal dialysis
* Primary peritonitis
* Immunocompromised (ongoing chemotherapy or prednisolone >20 mg/day)
* Chronic parenchymal liver disease
* Pregnancy
* Patients with end-stage disease
* Laparoscopic surgery (not converted to laparotomy)
* Acute occlusion of superior mesenteric artery
* Peritoneal carcinomatosis
* Abdominal trauma
* Lack of consent from the surgical equipoise
* Local peritonitis confined to 1 quadrant only

Randomization

Patients are included by a surgical equipoise followed by patient information and consent after recovery. The primary investigator from each site will be contacted by the surgeon on-call when a patient is scheduled for diagnostic laparoscopy or explorative laparotomy on suspicion of secondary peritonitis. Patients' fulling inclusions criteria will be randomized after consent has been obtained by the surgical equipoise. Centers that do not receive approval from their respective scientific ethics committee to include patients through a surgical equipoise must obtain informed and written consent before randomization. Randomization will be web-based via (REDCap ®) in blocks of 2, 4, and 6 stratified for center and age above or below 65 years. The justifications for stratifying according to the center are that there might be differences in the surgical treatment, preoperative optimization, and postoperative treatment both at the ward and intensive care unit (ICU) that might affect the outcome. The patients will be randomized to either abdominal closure with ROD or open abdomen with VAC. The randomization tool, along with eligibility criteria, can be accessed through our website, www.vacor.sdu.dk.

In cases where the surgeon finds that the allocated treatment may be contraindicated or is judged to harm the patient, it will be left to the surgeon's discretion to choose the most appropriate treatment. Patients who cannot be treated according to randomization will be analyzed according to intention-to-treat principles. Any eligible patient not included will be registered in a screening log.

How to apply Vacuum Assisted Closure (VAC)

The VAC® Abdominal Dressing System (KCI Vacuum Assisted Closure, San Antonio, TX, USA) will be used. Intestines, including lateral aspects, are covered by the visceral protective layer. The first layer of foam is placed in the laparostoma on the visceral protective layer and must extend below the fascia at a distance of 5 cm from the facial opening. Above this, a minimum of one piece of foam is folded and placed in the laparostoma. Finally, the laparostoma will be covered by the occlusive drape. A circular opening of approximately 5 cm in diameter will be created in the drape where the connection tubes to the vacuum pump will be placed. Simultaneously while applying the negative pressure of 125 mmHg, the wound edges are approximated manually towards the midline. The dressing will be changed with an interval of approximately 48 hours as standard or whenever needed according to the clinical condition. Each dressing change must be performed in the operation theatre with the patient in general anesthesia and muscle relaxation. Peritoneal fluid must be cultured at each dressing change and when fascia is closed. The fascia closure will commence as soon as possible according to the patient's general condition judged by gastrointestinal function, renal function, and a decline in inflammatory parameters either in one or repeated sessions. The aim will be a closure of the abdomen within a maximum of 8 days after the index operation.

The fascia closure after VAC-treatment can be according to the Israelssons principle as described below or upon the surgeon's discretion. A staged closure may start distally, proximally, or in a combination.

How to do primary closure

The abdominal wall is closed according to the Isreaelsson principle where it is sewn continuously in the fascia at a distance between the sutures of 5 mm and the distance to the facade edge of 5-10 mm. Monofilament PDS 0-0 (Ethicon) (or equivalent) is used. The suturing is started cranially and caudally, and the sutures are tied at the end of the continuous thread with self-locking knots. 4 times as much suture material as the length of the wound must be consumed.

The fascia closure after VAC-treatment can be according to the Israelssons principle as described below or upon the surgeon's discretion. A staged closure may start distally, proximally, or in a combination.

Postoperative course

Immediately after index operation, the surgeon fills out the baseline form containing patient characteristics and comorbidities, etiology of the peritonitis, surgical procedure, and the complexity of the condition according to Björck's classification. Patients can be transferred postoperatively to the intensive care unit (ICU) or the ward at the discretion of the treating team. Upon arrival to either the ward or the ICU, Acute Physiology and Chronic Health Evaluation II (APACHE II) and sequential organ failure assessment (SOFA) score must be performed by the attending anesthesiologist. SOFA-scoring and routine blood samples with CRP, bilirubin, creatinine, and platelets must be performed daily within the first seven days after index operation. Discharge from the ICU will be at the discretion of the attending intensivist and surgeon.

After completion of treatment

At hospital discharge, the patients will be booked for follow-up after 12 months in the outpatient clinic for abdominal palpation and abdominal CT-scan with intravenous contrast and Valsalva maneuver. In addition, the SF-36 questionnaire will be completed at 3- and 12-months follow-up.

Power calculation

With an expected peritonitis related complications rate of 40% in the ROD group and 25% in the VAC group, the desired power of 80%, a significance level of 0.05, and an expected drop-out of 5% a total of 340 patients should be included. With this sample size a 0.32 standard deviation difference in mean CCI between the two groups could be detected with 80% as well.

To ensure sufficient recruitment, the study will be multicentre and European. Eight active centers have been included, and two are in process. Randomization tools along with eligibility criteria are accessible through our website. The workflow and relevant contact details appear on posters at the participating departments. Study progress will be available on the website.

Statistical analysis

Patient characteristics will be summarized with frequencies and proportions (for categorical variables) or with mean values ± standard deviation, median values, quartiles, and minimum and maximum values (for numerical variables). Categorical variables will be compared using a Fisher's exact test and continuous variables with a Wilcoxon rank-sum test.

The primary peritonitis-related complication outcome will be compared between intervention groups by chi-squared test, reported as relative risk with 95% CI. The CCI outcome will be compared by linear regression with bootstrapped standard errors reporting mean difference with 95% confidence intervals.

A superiority and a non-inferiority analysis VAC treatment against primary closure with ROD will be performed. Applying non-inferiority margin of 5% of the peritonitis related complications.

An univariate analysis will be performed on the individual complication types (abscess, leakage, etc.) and complications as a whole (peritonitis related complications and CCI). Fisher's exact or chi-square test will be used to compare the treatments depending on the number of observations.

Adjusted analysis by logistic regression will be performed for complications as a whole and for the individual complications as an outcome, where it will be adjusted for age, performance status, and comorbidity. The above analyses will also be performed as a subgroup analysis where patients with APACHE-II score> ten will be included. This evaluates VAC and ROD in the most seriously ill part of the patient population.

The hospital health care utility and average treatment costs are compared between the treatment groups. The resource use will be reported as the mean difference with 95% confidence intervals (CI) compared by linear regression. In case of deviations from normality assumptions, bootstrapping with 1000 repetitions will be performed. Finally, the proportion of patients who experience radiological, acute operations will be compared by binomial regression estimating relative risk (RR) with 95% CI.

The interim analysis will be performed at 25%, 50%, and 75% of recruited patients on the primary outcome after 30-days to detect significant differences between groups at the earliest possible time, ultimately leading to the termination of the study. We have adjusted our power calculation to the interim analyses using the O'Brian-Flemming method. The study group will have access to the results of the interim analyses and may make the final decision to terminate the study.

All of the above analyses will be performed as both intention-to-treat (patients will be analyzed according to their randomization group) and per-protocol analysis (what actually happened). The main analyses will be performed as complete case analyses. Multiple imputations will impute missing values in a supplementary analysis, including baseline characteristics as predictors.

P values less than 0.05 will be considered statistically significant. Statistical calculations will be performed using Stata software (version 15, Stata Corp LP, Texas, USA).

Ethics

The study will be conducted in accordance with the Declaration of Helsinki and complies with current GDPR recommendations. The regional Danish Medical Ethics committee has approved the study to include patients in the acute setting with temporary consent by a surgical equipoise followed by patient information and consent after recovery. The surgical equipoise must not have any personal interest in the experiment, have experience, or have knowledge about the disease and the risks and benefits of the treatments and be indifferent to the therapeutic value of the two interventions. The rationale for choosing this inclusion model was that the subjects require immediate surgical intervention, are partly or entirely incapable of receiving and understanding the information. The severity of the condition does not allow time for third-party authorization. Both treatment regimens are accepted, safe, and widely used for this patient group. After the convalescence, patients will be informed about the project, and consent will be obtained. In instances where the patients do not survive before regaining habitual state, surrogate consent will be obtained. The patient can withdraw from the experiment at any time without having to explain him- or herself.

Patients in Denmark are covered by national insurance (Patienterstatningen), international centers will use country-specific insurance regulations. The study is investigator-initiated without economic interest to manufacturers or others involved in the investigation. No financial resources will be provided to the trial participants. Participating centers will receive the amount of 4000 Danish Krone per included patient yearly to cover the CT-scan of the abdomen and follow-up at the outpatient clinic.

The final data set will be available to the project owner and data assessor. Data can be shared in an anonymized form after an approved agreement on request. The primary investigator is responsible for data collection and handling. Unexpected adverse events must be reported to the regional committee of ethics.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for enrolment are 18+ years of age and are scheduled for acute laparotomy due to suspected peritonitis originating from perforation of the small bowel, colon, or rectum. To be included, purulent, enteric, or fecal contamination in a minimum of 2 out of 4 quadrants must be confirmed.

Exclusion Criteria:

* Diffuse peritonitis originating from a different focus than the small intestine, colon or rectum
* Diffuse peritonitis originating from a perforation on the stomach, duodenum, gallbladder, appendix, necrotizing pancreatitis, salpingitis, or peritoneal dialysis
* Primary peritonitis
* Immunocompromised (ongoing chemotherapy or prednisolone >20 mg/day)
* Chronic parenchymal liver disease
* Pregnancy
* Patients with end-stage disease
* Laparoscopic surgery (not converted to laparotomy)
* Acute occlusion of superior mesenteric artery
* Peritoneal carcinomatosis
* Abdominal trauma
* Lack of consent from the surgical equipoise
* Local peritonitis confined to 1 quadrant only

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint is to compare peritonitis related complications and Comprehensive Complication Index (CCI) between NPWT treatment (VAC) and conventional treatment (ROD) at 30, 90 days and 1 year. | 1 year
  Disease-Related Major Morbidity Needing Readmission and Conservative Treatment but Not Surgery
  * Fistula
  * Wound dehiscence/incisional hernia with obstruction
  * Abscess needing percutaneous drainage
  * Renal failure
  * Myocardial infarction
  * Gastric or duodenal bleeding
  * Respiratory failure
  * Urosepsis
  Disease-Related Major Morbidity Needing Surgical Intervention During First Admission or Readmission
  * Incisional hernia
  * Bowel obstruction or herniation due to intra-abdominal adhesions
  * Burst abdomen
  * Abdominal compartment syndrome
  * Fistula
  * Intra-abdominal bleeding
  * Intra-abdominal hematoma needing surgical evacuation
  * Perforation of visceral organ confirmed at surgery
  * Anastomotic leakage
  * Ischemia or necrosis of a visceral organ
  * Enterostomy dysfunction due to prolapse, stenosis, or retraction
  * Gastric or duodenal ulcer bleeding needing intervention of any type

SECONDARY OUTCOMES:
Mortality at 30, 90 days and 1 year | 1 year
  Mortality
Quality of life after treatment | 3 and 12 months
  Quality of life is measured after 3 and 12 months by the short form health survey (SF-36) questionnaire.
  The scale measures overall health status.
  SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  Following eight sections are included: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health.
Ventral hernia rate | 3 and 12 months
  Ventral hernia after after 12 months assessed by clinical examination and abdominal CT-scan with intravenous contrast +/- Valsalva maneuvre.
Hospital care utility within three months after index surgery | Up to 12 weeks
  Three months after the index operation, a record review will be made to estimate the health care utility and includes surgeries, total hospital stay, admissions at the ICU, and radiological interventions

OTHER OUTCOMES:
Microdialysis | First 4 days afte index laparatomy
  The concentration of lactate, glycerol, pyruvate, glucose, and cytokines in the peritoneal fluid in a subgroup of 10 patients from each group measured by intraperitoneal microdialysis postoperative day 0-4
Inscional hernia | 3 years
  Incisional hernia rate after three years assessed by a retrospective review of patient records

CONTACTS AND LOCATIONS:
Overall Officials: Niels Qvist, Professor, Study Director — Surgical Department A, Odense University Hospital, Denmark; Uffe Tange Holst, M.D., Study Chair — Surgical Department A, Odense University Hospital, Denmark; Jens Michelsen, M.D., Study Chair — Anesthesiology department V, Odense University Hospital, Denmark; Palle Toft, Professor, Study Chair — Anesthesiology department V, Odense University Hospital, Denmark
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rajabaleyan P, Michelsen J, Tange Holst U, Moller S, Toft P, Luxhoi J, Buyukuslu M, Bohm AM, Borly L, Sandblom G, Kobborg M, Aagaard Poulsen K, Schou Love U, Ovesen S, Grant Solling C, Morch Sondergaard B, Lund Lomholt M, Ritz Moller D, Qvist N, Bremholm Ellebaek M; VACOR study group. Vacuum-assisted closure versus on-demand relaparotomy in patients with secondary peritonitis-the VACOR trial: protocol for a randomised controlled trial. World J Emerg Surg. 2022 May 26;17(1):25. doi: 10.1186/s13017-022-00427-x. PMID 35619144